CLINICAL TRIAL: NCT05145881
Title: Evaluation of Clinical Effect of Probiotics in Alzheimer's Disease: a Randomized, Double-blind Clinical Trial
Brief Title: Effect of Probiotics in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hsieh-Hsun Ho (Industry)
Responsible Party: Sponsor-Investigator, Hsieh-Hsun Ho, R&D Director, Glac Biotech Co., Ltd
Organization: Glac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECKIRB1080701
Record Dates: First submitted 2021-11-11; First posted 2021-12-06 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Intestinal flora; Probiotics; Gut microbiota-brain axis (GMBA)
MeSH Terms: conditions — Alzheimer Disease | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose probiotics (Active Comparator)
  Interventions: Dietary Supplement: Low dose probiotics
- Normal dose probiotics (Experimental)
  Interventions: Dietary Supplement: Normal dose probiotics

INTERVENTIONS:
Dietary Supplement: Low dose probiotics — Taking 1 package of low dose probiotic powder (B. breve Bv-889, B. longum subsp. infantis BLI-02, B. bifidum VDD088, B. animalis subsp. lactis CP-9, Lactobacillus plantarum PL-02) twice daily before meals (BIDAC).
  Arms: Low dose probiotics
Dietary Supplement: Normal dose probiotics — Taking 1 package of normal dose probiotic powder (B. breve Bv-889, B. longum subsp. infantis BLI-02, B. bifidum VDD088, B. animalis subsp. lactis CP-9, Lactobacillus plantarum PL-02) twice daily before meals (BIDAC).
  Arms: Normal dose probiotics

SUMMARY:
In this clinical trial, five strains of probiotics (Bifidobacterium breve Bv-889, B. longum subspecies infantis BLI-02, B. bifidum VDD088, B. animalis subsp. lactis CP-9, Lactobacillus plantarum PL-02) with anti-oxidant and anti-inflammatory functions will been applied to slow down the development of the Alzheimer's disease through regulating the intestinal flora and immune system of patients with mild to moderate Alzheimer's disease symptoms. The efficacy of probiotic treatment against Alzheimer's disease will be evaluated.

DETAILED DESCRIPTION:
Alzheimer's disease is a neurodegenerative disease that mainly results in dementia. According to statistics, about 60-70% of dementia patients in Taiwan are Alzheimer's patients. Currently, there is no effective medical treatments for Alzheimer's disease. Several drugs and psychotherapy have been developed to attenuate the symptoms of the disease. The initial symptoms of Alzheimer's disease are memory loss of recent events (short-term memory impairment) and the disease can eventually deprive the patient's self-awareness in the late phase. The main factor leading to Alzheimer's disease is rapid apoptosis of neuronal cells in the brain.

The neuronal apoptosis is mainly due to abnormal chronic inflammatory reactions and oxidative stress. The gut microbiota-brain axis (GMBA) reflects the two-way communication between the central nervous system (CNS) and the gastrointestinal tract. It has been reported that GMBA dysregulation is closely related to neurodegenerative diseases.

Elmira Akbari et al showed that patients with Alzheimer's disease supplemented with both Bifidobacterium and Lactobacillus for 12 weeks expressed significantly higher Mini-Mental State Examination (MMSE) scores than placebo group. Remarkably, biochemical indicators in the patient's serum, such as C-reactive protein and triglyceride were also improved significantly. However, the clinical study of Elmira Akbari did not further explore the role of Bifidobacterium in controlling Alzheimer's disease.

In this clinical trial, patients will be randomly divided into 2 groups: low dose probiotics and normal dose probiotics. All patients will be supplemented with the probiotics for 12 weeks. Their (1) cognitive function, (2) cognitive behavioral ability, (3) sleep status (4) cerebral blood flow (5) blood immune variation spectrum and blood biochemical indicators and (6) variation of fecal flora will be analyze. The therapeutic efficiency of the probiotics will be further evaluated by comparing the changes in data before and after probiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 50-95 years old.
* The subject is clinically diagnosed with Alzheimer's disease, and it meets the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDB) or National Institute on Aging and Alzheimer's Association (NIAAA).
* The subject's MMSE score is between 10-25.
* The subject's CDR score is 0.5, 1, or 2.
* The subject can cooperate to perform cognitive function tests.
* The subject who have dependable caregivers who can record the compliance of taking probiotics and any physical conditions.
* The subject or family members have signed the informed consent form.

Exclusion Criteria:

* The subject is shown to have cerebrovascular disease by computer tomography.
* The subject has dementia caused by other reasons, such as brain trauma, tumor, infection, epilepsy, etc.
* The subject has used immunosuppressant drugs, steroids, T cell inhibitor ointments or received chemotherapy within 2 weeks.
* The subject has consumed probiotic-related products (probiotic powder, yogurt or other fermented foods) within the past 1 month.
* The subject has participated in clinical trials of other dementia medications in the past 1 month.
* The subject is assessed for dementia caused by vitamin B12 deficiency or thyroid abnormalities.
* The subject suffers from mental illness, severe depression, schizophrenia, drug addiction, and alcohol addiction.
* The subject has Parkinson's disease.
* The subject is assessed to have severe metabolic dysfunction, liver and kidney dysfunction.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-COG) | At day 0 and 12th week.
  The minimum score is 0 and the maximum score is 70. A higher score means more severe cognitive impairment. The change in score before and after probiotic intervention will be evaluated.
Clinician's Interview-Based Impression of Severity (CIBIS) | At day 0.
  The minimum score is 1 and the maximum score is 7. A higher score means more severe mental illness. The change in score before and after probiotic intervention will be evaluated.
Clinician's Interview-Based Impression of Severity--plus caregiver input (CIBIS-plus) | At 12th week.
  The minimum score is 1 and the maximum score is 7. A higher score means more severe mental illness. The change in score before and after probiotic intervention will be evaluated.

SECONDARY OUTCOMES:
Cognitive behavioral ability | At day 0 and 12th week.
  Evaluating the score difference of the following 3 indicators before and after probiotic intervention:
  1. Mini-Mental State Examination (MMSE). The minimum score is 0 and the maximum score is 30. A higher score means better cognitive function.
  2. Clinical Dementia Rating (CDR). The minimum score is 0 and the maximum score is 3. A higher score means more severe dementia.
  3. Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL). The minimum score is 0 and the maximum score is 54. A higher score means better activities of daily living.
The length of the sleep period | At day 0 and 12th week.
  Wrist activity monitors will be used to record the length of the sleep period (hours) before and after the probiotic intervention.
The length of wake up after falling asleep | At day 0 and 12th week.
  Wrist activity monitors will be used to record the length of wake up (hours) after falling asleep before and after the probiotic intervention.
The total sleep time on the bed | At day 0 and 12th week.
  Wrist activity monitors will be used to record the total sleep time (hours) on the bed before and after the probiotic intervention.
Sleep efficiency | At day 0 and 12th week.
  Calculating sleep efficiency based on the length of the sleep period and the total sleep time on the bed recorded by Wrist activity monitors. [(Sleep efficiency = The length of the sleep period/The total sleep time on the bed)*100%]
Cerebral blood flow | At day 0 and 12th week.
  Using single photon emission computed tomography (SPECT/CT) to evaluate the changes in cerebral blood flow before and after probiotic intervention.
Blood immune variation spectrum and blood biochemical indicators. | At day 0 and 12th week.
  1. Detecting the changes of concentration in blood biochemical indexes, oxidative stress and cytokines before and after probiotic intervention.
  2. Detecting the changes of blood RNA level in the immune profile of IgG and IgA before and after the intervention of probiotics.
Fecal flora | At day 0 and 12th week.
  Using Next-Generation Sequencing (NGS) to analyze the changes of fecal flora before and after probiotic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hsieh-Hsun Ho, Ph.D, Principal Investigator — Glac Biotech Co., Ltd
Locations (1):
- Glac Biotech Co., Ltd, Tainan, Taiwan